CLINICAL TRIAL: NCT05396287
Title: The Impact of Cerebral Anatomical Variations on Cerebrovascular Reactivity
Brief Title: Blood Vessel Anatomy and Blood Flow Regulation
Status: Active, not recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0423; 1RF1NS117746-01 (NIH); Protocol Version 4/6/2022 (Other: UW Madison); A176000 (Other: UW Madison)
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Brain Blood Flow; Healthy
Keywords: MRI; Brain blood flow

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum blood samples will be retained for future analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Controls: Healthy controls
  Interventions: Device: MRI
- Vertebral Artery Hypoplasia: Healthy individuals with vertebral artery hypoplasia
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Participants will undergo an MRI scan while participating in two breathing tests (hypercapnia and hypoxia) to measure brain blood flow.

SUMMARY:
Brain blood flow regulation will be measured in response to environmental changes using MRI.

DETAILED DESCRIPTION:
Global brain blood flow decreases with advancing age; however, some adults have accelerated declines in brain blood flow, placing them at a greater risk of cognitive impairment. Similarly, brain reactivity to increased levels of carbon dioxide decreases with age, with a greater decline in adults with vascular risk factors and is impaired in early Alzheimer's disease. Preclinical models suggest that reduced brain blood flow, results in low levels of oxygen regionally. Currently, there are a lack of human studies that investigate the cause or consequence of altered blood flow regulation in the brain.

The research aims are:

1. Determine the impact of vertebral artery hypoplasia (VAH) on brain reactivity to increased levels of carbon dioxide.
2. Determine the impact of VAH on the brain blood flow response to acute low levels of oxygen.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≤38.5 kg/m2
* Nonsmoker
* Female subjects: postmenopausal
* Currently enrolled in the Wisconsin Alzheimer's Disease Research Clinical Core

Exclusion Criteria:

* Diagnosis of mild cognitive impairment or Alzheimer's disease
* Uncontrolled hypertension
* History or evidence of hepatic disease, hematological disease, or peripheral vascular disease
* Severe kidney injury requiring hemodialysis
* Cardiovascular disease including: severe congestive heart failure, coronary artery disease, ischemic heart disease (stents, coronary artery bypass grafts) and tachycardia
* History of clinically significant ischemic or hemorrhagic stroke, or significant cerebrovascular disease
* History of HIV/AIDS
* Severe untreated obstructive sleep apnea
* History of diabetes with HbA1c greater than 9.5%
* Major neurologic disorders other than dementia (e.g., multiple sclerosis, amyotrophic lateral sclerosis, brain surgery, etc.)
* Current or recent (<1 year) major psychiatric condition (Axis I) or addictive disorders
* Contraindications to MRI

Ages: 55 Years to 69 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects for this study, will include healthy adults enrolled in the Wisconsin Alzheimer's Disease Research Clinical Core. Both men and women are eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Cerebral Vascular Reactivity to Hypercapnia | One study visit, up to 120 minutes in the MRI
  The change in brain blood flow using MRI will be measured in response to a hypercapnic breathing test. The participants cerebral vascular reactivity to hypercapnia will be compared between the controls (without VAH) and those with VAH.
Cerebral Blood Flow Response to Hypoxia | One study visit, up to 120 minutes in the MRI
  The change in brain blood flow using MRI will be measured in response to a hypoxic breathing test. The participants cerebral blood flow response to hypoxia will be compared between the controls (without VAH) and those with VAH.

CONTACTS AND LOCATIONS:
Overall Officials: Jill N Barnes, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kisler K, Nelson AR, Montagne A, Zlokovic BV. Cerebral blood flow regulation and neurovascular dysfunction in Alzheimer disease. Nat Rev Neurosci. 2017 Jul;18(7):419-434. doi: 10.1038/nrn.2017.48. Epub 2017 May 18. PMID 28515434
- [Background] Switzer AR, Cheema I, McCreary CR, Zwiers A, Charlton A, Alvarez-Veronesi A, Sekhon R, Zerna C, Stafford RB, Frayne R, Goodyear BG, Smith EE. Cerebrovascular reactivity in cerebral amyloid angiopathy, Alzheimer disease, and mild cognitive impairment. Neurology. 2020 Sep 8;95(10):e1333-e1340. doi: 10.1212/WNL.0000000000010201. Epub 2020 Jul 8. PMID 32641520
- [Background] Iadecola C. Neurovascular regulation in the normal brain and in Alzheimer's disease. Nat Rev Neurosci. 2004 May;5(5):347-60. doi: 10.1038/nrn1387. No abstract available. PMID 15100718
- [Background] Scheel P, Puls I, Becker G, Schoning M. Volume reduction in cerebral blood flow in patients with vascular dementia. Lancet. 1999 Dec 18-25;354(9196):2137. doi: 10.1016/S0140-6736(99)04016-7. PMID 10609827
- [Background] Marshall RS, Lazar RM. Pumps, aqueducts, and drought management: vascular physiology in vascular cognitive impairment. Stroke. 2011 Jan;42(1):221-6. doi: 10.1161/STROKEAHA.110.595645. Epub 2010 Dec 9. PMID 21148438
- [Background] Wierenga CE, Hays CC, Zlatar ZZ. Cerebral blood flow measured by arterial spin labeling MRI as a preclinical marker of Alzheimer's disease. J Alzheimers Dis. 2014;42 Suppl 4(Suppl 4):S411-9. doi: 10.3233/JAD-141467. PMID 25159672
- [Background] Park JH, Kim JM, Roh JK. Hypoplastic vertebral artery: frequency and associations with ischaemic stroke territory. J Neurol Neurosurg Psychiatry. 2007 Sep;78(9):954-8. doi: 10.1136/jnnp.2006.105767. Epub 2006 Nov 10. PMID 17098838
- [Background] Thierfelder KM, Baumann AB, Sommer WH, Armbruster M, Opherk C, Janssen H, Reiser MF, Straube A, von Baumgarten L. Vertebral artery hypoplasia: frequency and effect on cerebellar blood flow characteristics. Stroke. 2014 May;45(5):1363-8. doi: 10.1161/STROKEAHA.113.004188. Epub 2014 Apr 3. PMID 24699051
- [Background] Peterson C, Phillips L, Linden A, Hsu W. Vertebral artery hypoplasia: prevalence and reliability of identifying and grading its severity on magnetic resonance imaging scans. J Manipulative Physiol Ther. 2010 Mar-Apr;33(3):207-11. doi: 10.1016/j.jmpt.2010.01.012. PMID 20350674
- [Background] Kulyk C, Voltan C, Simonetto M, Palmieri A, Farina F, Vodret F, Viaro F, Baracchini C. Vertebral artery hypoplasia: an innocent lamb or a disguise? J Neurol. 2018 Oct;265(10):2346-2352. doi: 10.1007/s00415-018-9004-7. Epub 2018 Aug 16. PMID 30116939
- [Background] Chen G, Ward BD, Xie C, Li W, Wu Z, Jones JL, Franczak M, Antuono P, Li SJ. Classification of Alzheimer disease, mild cognitive impairment, and normal cognitive status with large-scale network analysis based on resting-state functional MR imaging. Radiology. 2011 Apr;259(1):213-21. doi: 10.1148/radiol.10100734. Epub 2011 Jan 19. PMID 21248238
- [Background] Bangen KJ, Nation DA, Clark LR, Harmell AL, Wierenga CE, Dev SI, Delano-Wood L, Zlatar ZZ, Salmon DP, Liu TT, Bondi MW. Interactive effects of vascular risk burden and advanced age on cerebral blood flow. Front Aging Neurosci. 2014 Jul 7;6:159. doi: 10.3389/fnagi.2014.00159. eCollection 2014. PMID 25071567
- [Background] Barnes JN, Schmidt JE, Nicholson WT, Joyner MJ. Cyclooxygenase inhibition abolishes age-related differences in cerebral vasodilator responses to hypercapnia. J Appl Physiol (1985). 2012 Jun;112(11):1884-90. doi: 10.1152/japplphysiol.01270.2011. Epub 2012 Mar 22. PMID 22442028
- [Background] Barnes JN, Harvey RE, Miller KB, Jayachandran M, Malterer KR, Lahr BD, Bailey KR, Joyner MJ, Miller VM. Cerebrovascular Reactivity and Vascular Activation in Postmenopausal Women With Histories of Preeclampsia. Hypertension. 2018 Jan;71(1):110-117. doi: 10.1161/HYPERTENSIONAHA.117.10248. Epub 2017 Nov 20. PMID 29158356
- [Background] Tchistiakova E, Crane DE, Mikulis DJ, Anderson ND, Greenwood CE, Black SE, MacIntosh BJ. Vascular risk factor burden correlates with cerebrovascular reactivity but not resting state coactivation in the default mode network. J Magn Reson Imaging. 2015 Nov;42(5):1369-76. doi: 10.1002/jmri.24917. Epub 2015 Apr 17. PMID 25884110
- [Background] Alwatban M, Murman DL, Bashford G. Cerebrovascular Reactivity Impairment in Preclinical Alzheimer's Disease. J Neuroimaging. 2019 Jul;29(4):493-498. doi: 10.1111/jon.12606. Epub 2019 Feb 12. PMID 30748053
- [Background] Moskowitz MA, Lo EH, Iadecola C. The science of stroke: mechanisms in search of treatments. Neuron. 2010 Jul 29;67(2):181-98. doi: 10.1016/j.neuron.2010.07.002. PMID 20670828
- [Background] Wong SM, Jansen JFA, Zhang CE, Hoff EI, Staals J, van Oostenbrugge RJ, Backes WH. Blood-brain barrier impairment and hypoperfusion are linked in cerebral small vessel disease. Neurology. 2019 Apr 9;92(15):e1669-e1677. doi: 10.1212/WNL.0000000000007263. Epub 2019 Mar 13. PMID 30867275
- [Background] Peng SL, Chen X, Li Y, Rodrigue KM, Park DC, Lu H. Age-related changes in cerebrovascular reactivity and their relationship to cognition: A four-year longitudinal study. Neuroimage. 2018 Jul 1;174:257-262. doi: 10.1016/j.neuroimage.2018.03.033. Epub 2018 Mar 19. PMID 29567504
- [Background] Miller KB, Howery AJ, Rivera-Rivera LA, Johnson SC, Rowley HA, Wieben O, Barnes JN. Age-Related Reductions in Cerebrovascular Reactivity Using 4D Flow MRI. Front Aging Neurosci. 2019 Oct 17;11:281. doi: 10.3389/fnagi.2019.00281. eCollection 2019. PMID 31680935
- [Background] Iqbal S. A comprehensive study of the anatomical variations of the circle of willis in adult human brains. J Clin Diagn Res. 2013 Nov;7(11):2423-7. doi: 10.7860/JCDR/2013/6580.3563. Epub 2013 Nov 10. PMID 24392362
- [Background] Hays CC, Zlatar ZZ, Wierenga CE. The Utility of Cerebral Blood Flow as a Biomarker of Preclinical Alzheimer's Disease. Cell Mol Neurobiol. 2016 Mar;36(2):167-79. doi: 10.1007/s10571-015-0261-z. Epub 2016 Feb 22. PMID 26898552
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Slessarev M, Han J, Mardimae A, Prisman E, Preiss D, Volgyesi G, Ansel C, Duffin J, Fisher JA. Prospective targeting and control of end-tidal CO2 and O2 concentrations. J Physiol. 2007 Jun 15;581(Pt 3):1207-19. doi: 10.1113/jphysiol.2007.129395. Epub 2007 Apr 19. PMID 17446225
- [Background] Poublanc J, Sobczyk O, Shafi R, Sayin ES, Schulman J, Duffin J, Uludag K, Wood JC, Vu C, Dharmakumar R, Fisher JA, Mikulis DJ. Perfusion MRI using endogenous deoxyhemoglobin as a contrast agent: Preliminary data. Magn Reson Med. 2021 Dec;86(6):3012-3021. doi: 10.1002/mrm.28974. Epub 2021 Oct 22. PMID 34687064
- [Background] Mikhail Kellawan J, Harrell JW, Roldan-Alzate A, Wieben O, Schrage WG. Regional hypoxic cerebral vasodilation facilitated by diameter changes primarily in anterior versus posterior circulation. J Cereb Blood Flow Metab. 2017 Jun;37(6):2025-2034. doi: 10.1177/0271678X16659497. Epub 2016 Jan 1. PMID 27406213
- [Background] Barton GP, Corrado PA, Francois CJ, Chesler NC, Eldridge MW, Wieben O, Goss KN. Exaggerated Cardiac Contractile Response to Hypoxia in Adults Born Preterm. J Clin Med. 2021 Mar 10;10(6):1166. doi: 10.3390/jcm10061166. PMID 33802149
- [Background] Mardimae A, Balaban DY, Machina MA, Battisti-Charbonney A, Han JS, Katznelson R, Minkovich LL, Fedorko L, Murphy PM, Wasowicz M, Naughton F, Meineri M, Fisher JA, Duffin J. The interaction of carbon dioxide and hypoxia in the control of cerebral blood flow. Pflugers Arch. 2012 Oct;464(4):345-51. doi: 10.1007/s00424-012-1148-1. Epub 2012 Sep 9. PMID 22961068
- [Background] Miller KB, Howery AJ, Harvey RE, Eldridge MW, Barnes JN. Cerebrovascular Reactivity and Central Arterial Stiffness in Habitually Exercising Healthy Adults. Front Physiol. 2018 Aug 17;9:1096. doi: 10.3389/fphys.2018.01096. eCollection 2018. PMID 30174609
- [Background] Barnes JN, Harvey RE, Eisenmann NA, Miller KB, Johnson MC, Kruse SM, Lahr BD, Joyner MJ, Miller VM. Cerebrovascular reactivity after cessation of menopausal hormone treatment. Climacteric. 2019 Apr;22(2):182-189. doi: 10.1080/13697137.2018.1538340. Epub 2019 Jan 21. PMID 30661405
- [Background] Ahmed M, Giesbrecht GG, Serrette C, Georgopoulos D, Anthonisen NR. Ventilatory response to hypoxia in elderly humans. Respir Physiol. 1991 Mar;83(3):343-51. doi: 10.1016/0034-5687(91)90053-l. PMID 2052762
- [Background] Vovk A, Smith WD, Paterson ND, Cunningham DA, Paterson DH. Peripheral chemoreceptor control of ventilation following sustained hypoxia in young and older adult humans. Exp Physiol. 2004 Nov;89(6):647-56. doi: 10.1113/expphysiol.2004.027532. Epub 2004 Jul 15. PMID 15258116